CLINICAL TRIAL: NCT02745847
Title: The Safety and Efficacy of Re-irradiation With Stereotactic Body Radiotherapy for Relapsed Pancreatic Cancer
Brief Title: Re-irradiation With Stereotactic Body Radiotherapy for Relapsed Pancreatic Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhang Huo Jun, Director of Radiation Oncology Department, Changhai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChangH Hosp
Record Dates: First submitted 2016-04-15; First posted 2016-04-20 (Estimated); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Re-Irradiation; Radiosurgery

STUDY DESIGN:
Intervention Model Description: Re-irradiation with SBRT
Oversight: Data Monitoring Committee: No

ARMS (1):
- Re-irradiation with SBRT (Experimental): Patients with relapsed pancreatic cancer meeting all inclusion criteria will receive re-irradiation with SBRT.
  Interventions: Radiation: Re-irradiation with SBRT

INTERVENTIONS:
Radiation: Re-irradiation with SBRT — Patients previously treated with SBRT with relapsed pancreatic cancer will be re-irradiated with SBRT.

SUMMARY:
The safety and efficacy of re-irradiation with stereotactic body radiotherapy for relapsed pancreatic cancer will be evaluated.

DETAILED DESCRIPTION:
Pancreatic cancer is one of the most lethal malignant tumors, probably attributable to local recurrence deemed as a predominant factor influencing patients' prognosis and quality of life. Only 15%-20% patients are suitable for surgeries among those first diagnosed with pancreatic cancer and the 5-year survival rate of those patients with R0 resection is still less than 20%. Therefore, radiotherapy is becoming a promising method to improve survival. However, due to adjacent organs at risk, conventional external beam radiotherapy, besides long courses, sometimes results in severe radiation-induced toxicity, delaying the initial of thereafter treatment, such as chemotherapy, which reduces clinical benefits.

A single-fraction dose in the gross tumor volume could be increased stereotactic body radiotherapy (SBRT). Furthermore, doses of organs at risk could also be reduced, thus effectively improving local control rates and reducing radiation related toxicity. Compared with conventional external beam radiotherapy, SBRT is proved to provide longer progression free survival and safe with combination of chemotherapy. Moreover, owing to short courses and low toxicity of SBRT, quality of life is largely improved.

However, it was reported that progression usually occurred 2 years after the initial treatment. The most common failure pattern was local recurrence. Chemotherapy and supportive treatment were commonly used in relapsed pancreatic cancer but with unfavored outcomes. Palliative surgeries are performed in patients with recurrent pancreatic cancer in some studies. Nevertheless, because of bad medical conditions and high complication rates, many patients could not endure surgeries. Therefore, whether patients previously treated with SBRT could be re-irradiated is another challenge in the treatment of pancreatic cancer.

Some studies have confirmed that improved quality of life and longer survival could be available with re-irradiation via SBRT in patients with relapsed pancreatic cancer. Real-time guiding and synchronous tracing of SBRT increase the doses of tumor volumes but decrease doses of organs at risk and toxicity, rendering SBRT as an alternative treatment for relapsed pancreatic cancer. Chris et al. demonstrated that 1-year local control rate was 70% after re-irradiation with SBRT in 14 patients and the toxicity was mild. Nergiz Dagoglu et al. showed that the median overall survival was 14 months and no grade 3, 4 and 5 toxicities occurred.

From 2013-2015, we retrospectively reviewed medical records of 14 patients with relapsed pancreatic cancer re-irradiated with SBRT. All of their tumor markers and pain scores decreased and quality of life improved 3 months after re-irradiation. Hence, based on our experience, we attempt to prospectively evaluate the safety and efficacy of re-irradiation with SBRT for relapsed pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18
2. KPS≥70
3. Pancreatic malignancy need to be confirmed by histological or cytological valuation or clinical diagnosis (MDT with typical clinical manifestations, radiological features of pancreatic cancer via MRI and PET-CT).
4. Patients were previously treated with SBRT in Shanghai Changhai hospital
5. The time from the end of prior SBRT to local recurrence is more than 6 months
6. In-field recurrences of pancreatic cancer confirmed by Imaging examinations.
7. Blood routine examination: Absolute neutrophil count (ANC) ≥ 1.5 ×10^9/L, leukocyte count≥ 3.5 ×10^9/L, platelets ≥ 70×10^9/L, hemoglobin ≥ 80 g/L
8. Blood routine examination: Absolute neutrophil count (ANC) ≥ 1.5 ×10^9/L, leukocyte count≥ 3.5 ×10^9/L, platelets ≥ 70×10^9/L, hemoglobin ≥ 80 g/L
9. INR < 2 (0.9-1.1), PPT <1.5 × ULN
10. Ability of the research subject or authorized legal representative to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Age<18
2. KPS<70
3. Prior anti-tumor treatment (surgery, chemotherapy, radiation etc.) for the relapsed pancreatic cancer.
4. Evidences of metastatic disease or invasion of the stomach or duodenum confirmed by Imaging examinations.
5. The time from the end of prior SBRT to local recurrence is less than 6 months
6. Patients with active inflammatory bowel diseases or peptic ulcer
7. Gastrointestinal bleeding or perforation within 6 months
8. Abnormal results of blood routine examinations and liver and kidney tests
9. Female who is pregnant or nursing, or is of childbearing potential and not using a reliable method of contraception
10. Patients with a history of any other malignancy (except basal cell carcinoma and carcinoma in situ of cervix)
11. Contraindication to SBRT
12. Inability of the research subject or authorized legal representative to understand and the willingness to sign a written informed consent document

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The toxicities following SBRT will be determined. | 3 years
  The toxicities following SBRT will be assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Overall survival | 3 years
  The median survival time will be determined.
Local recurrence-free survival | 3 years
  The local recurrence-free survival will be determined.
Objective response rates | 3 years
  The rate is the ratio of the number of patients with complete remission and partial remission to the total number of enrolled patients.
The quality of life will be analyzed. | 3 years
  The analysis of quality of life is based on QLQ-C30.
The quality of life will be analyzed. | 3 years
  The analysis of quality of life is based on QLQ-PAN26.

CONTACTS AND LOCATIONS:
Overall Officials: Huo Jun Zhang, MD., PH.D, Principal Investigator — Changhai Hospital
Locations (1):
- Huojun Zhang, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Tseng JF, Raut CP, Lee JE, Pisters PW, Vauthey JN, Abdalla EK, Gomez HF, Sun CC, Crane CH, Wolff RA, Evans DB. Pancreaticoduodenectomy with vascular resection: margin status and survival duration. J Gastrointest Surg. 2004 Dec;8(8):935-49; discussion 949-50. doi: 10.1016/j.gassur.2004.09.046. PMID 15585381
- [Background] Sener SF, Fremgen A, Menck HR, Winchester DP. Pancreatic cancer: a report of treatment and survival trends for 100,313 patients diagnosed from 1985-1995, using the National Cancer Database. J Am Coll Surg. 1999 Jul;189(1):1-7. doi: 10.1016/s1072-7515(99)00075-7. PMID 10401733
- [Background] HUGUET F H P V D. Impact of chemoradiation on local control and time without treatment in patients with locally advanced pancreatic cancer included in the international phase III LAP 07 study. Journal of Clinical Oncology 5s(32): 4001, 2014.
- [Background] Moningi S, Marciscano AE, Rosati LM, Ng SK, Teboh Forbang R, Jackson J, Chang DT, Koong AC, Herman JM. Stereotactic body radiation therapy in pancreatic cancer: the new frontier. Expert Rev Anticancer Ther. 2014 Dec;14(12):1461-75. doi: 10.1586/14737140.2014.952286. Epub 2014 Sep 3. PMID 25183386
- [Background] Berber B, Sanabria JR, Braun K, Yao M, Ellis RJ, Kunos CA, Sohn J, Machtay M, Teh BS, Huang Z, Mayr NA, Lo SS. Emerging role of stereotactic body radiotherapy in the treatment of pancreatic cancer. Expert Rev Anticancer Ther. 2013 Apr;13(4):481-7. doi: 10.1586/era.13.19. PMID 23560842
- [Background] Yechieli RL, Robbins JR, Mahan M, Siddiqui F, Ajlouni M. Stereotactic Body Radiotherapy for Elderly Patients With Medically Inoperable Pancreatic Cancer. Am J Clin Oncol. 2017 Feb;40(1):22-26. doi: 10.1097/COC.0000000000000090. PMID 24879474
- [Background] Kim CH, Ling DC, Wegner RE, Flickinger JC, Heron DE, Zeh H, Moser AJ, Burton SA. Stereotactic body radiotherapy in the treatment of pancreatic adenocarcinoma in elderly patients. Radiat Oncol. 2013 Oct 16;8:240. doi: 10.1186/1748-717X-8-240. PMID 24131503
- [Background] Rwigema JC, Parikh SD, Heron DE, Howell M, Zeh H, Moser AJ, Bahary N, Quinn A, Burton SA. Stereotactic body radiotherapy in the treatment of advanced adenocarcinoma of the pancreas. Am J Clin Oncol. 2011 Feb;34(1):63-9. doi: 10.1097/COC.0b013e3181d270b4. PMID 20308870
- [Background] Gurka MK, Collins SP, Slack R, Tse G, Charabaty A, Ley L, Berzcel L, Lei S, Suy S, Haddad N, Jha R, Johnson CD, Jackson P, Marshall JL, Pishvaian MJ. Stereotactic body radiation therapy with concurrent full-dose gemcitabine for locally advanced pancreatic cancer: a pilot trial demonstrating safety. Radiat Oncol. 2013 Mar 1;8:44. doi: 10.1186/1748-717X-8-44. PMID 23452509
- [Background] Mahadevan A, Miksad R, Goldstein M, Sullivan R, Bullock A, Buchbinder E, Pleskow D, Sawhney M, Kent T, Vollmer C, Callery M. Induction gemcitabine and stereotactic body radiotherapy for locally advanced nonmetastatic pancreas cancer. Int J Radiat Oncol Biol Phys. 2011 Nov 15;81(4):e615-22. doi: 10.1016/j.ijrobp.2011.04.045. Epub 2011 Jun 12. PMID 21658854
- [Background] Mukherjee S, Hurt CN, Bridgewater J, Falk S, Cummins S, Wasan H, Crosby T, Jephcott C, Roy R, Radhakrishna G, McDonald A, Ray R, Joseph G, Staffurth J, Abrams RA, Griffiths G, Maughan T. Gemcitabine-based or capecitabine-based chemoradiotherapy for locally advanced pancreatic cancer (SCALOP): a multicentre, randomised, phase 2 trial. Lancet Oncol. 2013 Apr;14(4):317-26. doi: 10.1016/S1470-2045(13)70021-4. Epub 2013 Mar 6. PMID 23474363
- [Background] Taniguchi CM, Murphy JD, Eclov N, Atwood TF, Kielar KN, Christman-Skieller C, Mok E, Xing L, Koong AC, Chang DT. Dosimetric analysis of organs at risk during expiratory gating in stereotactic body radiation therapy for pancreatic cancer. Int J Radiat Oncol Biol Phys. 2013 Mar 15;85(4):1090-5. doi: 10.1016/j.ijrobp.2012.07.2366. Epub 2012 Dec 27. PMID 23273994
- [Background] Sperti C, Moletta L, Merigliano S. Multimodality treatment of recurrent pancreatic cancer: Mith or reality? World J Gastrointest Oncol. 2015 Dec 15;7(12):375-82. doi: 10.4251/wjgo.v7.i12.375. PMID 26689800
- [Background] Miyazaki M, Yoshitomi H, Shimizu H, Ohtsuka M, Yoshidome H, Furukawa K, Takayasiki T, Kuboki S, Okamura D, Suzuki D, Nakajima M. Repeat pancreatectomy for pancreatic ductal cancer recurrence in the remnant pancreas after initial pancreatectomy: is it worthwhile? Surgery. 2014 Jan;155(1):58-66. doi: 10.1016/j.surg.2013.06.050. Epub 2013 Nov 12. PMID 24238124
- [Background] Lominska CE, Unger K, Nasr NM, Haddad N, Gagnon G. Stereotactic body radiation therapy for reirradiation of localized adenocarcinoma of the pancreas. Radiat Oncol. 2012 May 18;7:74. doi: 10.1186/1748-717X-7-74. PMID 22607687
- [Background] Dagoglu N, Callery M, Moser J, Tseng J, Kent T, Bullock A, Miksad R, Mancias JD, Mahadevan A. Stereotactic Body Radiotherapy (SBRT) Reirradiation for Recurrent Pancreas Cancer. J Cancer. 2016 Jan 10;7(3):283-8. doi: 10.7150/jca.13295. eCollection 2016. PMID 26918041
- [Background] Grimm J, LaCouture T, Croce R, Yeo I, Zhu Y, Xue J. Dose tolerance limits and dose volume histogram evaluation for stereotactic body radiotherapy. J Appl Clin Med Phys. 2011 Feb 8;12(2):3368. doi: 10.1120/jacmp.v12i2.3368. PMID 21587185
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Fitzsimmons D, Johnson CD, George S, Payne S, Sandberg AA, Bassi C, Beger HG, Birk D, Buchler MW, Dervenis C, Fernandez Cruz L, Friess H, Grahm AL, Jeekel J, Laugier R, Meyer D, Singer MW, Tihanyi T. Development of a disease specific quality of life (QoL) questionnaire module to supplement the EORTC core cancer QoL questionnaire, the QLQ-C30 in patients with pancreatic cancer. EORTC Study Group on Quality of Life. Eur J Cancer. 1999 Jun;35(6):939-41. doi: 10.1016/s0959-8049(99)00047-7. PMID 10533475